CLINICAL TRIAL: NCT06061484
Title: Safety Efficacy, and Cost-effectiveness of Modified Doses of Ready-to-use Therapeutic Food for the Treatment of Severe Acute Malnutrition Among Children 6-59 Months of Age in Ethiopia
Brief Title: Modified Dosage for Severe Acute Malnutrition
Acronym: MODAM-SAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Action Against Hunger USA (Other)
Collaborators: University of Washington (Other); Ethiopian Public Health Institute (Other Government)
Responsible Party: Principal Investigator, Heather Stobaugh, Senior Research and Learning Specialist, Action Against Hunger USA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MODAM-SAM
Record Dates: First submitted 2023-09-08; First posted 2023-09-29 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Standard weight-based dosing of Ready-to-Use Therapeutic Food (RUTF) at a dose of 150-200 kcal/kg/day
  Interventions: Dietary Supplement: ready-to-use therapeutic food (RUTF); Drug: Amoxicillin
- SAM Experimental A (Experimental): 2 sachets (1000 kcal) of RUTF per day
  Interventions: Dietary Supplement: ready-to-use therapeutic food (RUTF); Drug: Amoxicillin
- SAM Experimental B (Experimental): 2 sachets (1000 kcal) per day while MUAC < 115mm and/or edema and/or WHZ < -3; then decreasing to 1 sachet (500 kcal) per day while MUAC 115-124 and WHZ -2 to -3 and no edema
  Interventions: Dietary Supplement: ready-to-use therapeutic food (RUTF); Drug: Amoxicillin

INTERVENTIONS:
Dietary Supplement: ready-to-use therapeutic food (RUTF) — Standard formulation meeting UNICEF specifications: https://www.unicef.org/supply/sites/unicef.org.supply/files/2023-04/U239977-RUTF-Novel-Specification.pdf
Drug: Amoxicillin — Standard weight-based dosing per Ehtiopian national guidelines

SUMMARY:
Protocols for the community-based management of acute malnutrition (CMAM) have not changed significantly for more than 20 years, with relatively complex treatment protocols and persistent supply chain challenges that have limited overall program coverage, leaving millions of malnourished children without care annually. The overarching goal of this research project is to simultaneously test two novel simplified approaches in CMAM with potential to improve program coverage. The simplified approach includes two parallel clinical trials for SAM and MAM treatment. Two fixed-dose regimes of RUTF will be tested against the current weight-based dosing of RUTF for children with SAM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-59 months
2. Reside in the catchment area of the health post where the trial is to be conducted without plans to leave the area over the next year
3. Uncomplicated severe acute malnutrition, as defined by no signs of severe illness that would require referral to inpatient facility
4. Pass appetite test conducted at the time of enrollment
5. Consent for randomization into the study given by mother, father, and/or other primary caregiver
6. Mid-upper arm circumference less than 115 mm and/or nutritional edema
7. Weight-for-height Z-score (WHZ) less than -3

Exclusion Criteria:

1. Complicated acute malnutrition with severe illness requiring transfer to a stabilization center or hospital for treatment. This includes, but is not limited to: a. Hypothermia b. High fever c. Signs of hypoglycemia d. Lethargy or altered mental status e. Moderate to severe dehydration f. Shock g. Other medical complications requiring hospitalization or higher-level medical evaluation
2. Treatment for acute malnutrition, either as an inpatient or outpatient, within the past 3 months
3. Known chronic medical illness such as severe cerebral palsy, severe congenital anomalies such as unrepaired congenital heart disease, Down syndrome, hydrocephalus, unrepaired cleft lip or palate, or other conditions that would be expected to contribute to difficulty feeding the prescribed amounts of therapeutic or supplementary food

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2400 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
short-term nutritional recovery from severe acute malnutrition (SAM) | up to 16 weeks
  two consecutive weeks with MUAC > 12.4 cm and/or WHZ >= -2 and/or resolution of edema, depending on enrollment criteria

SECONDARY OUTCOMES:
weight gain during treatment | weekly for up to 16 weeks
MUAC gain during treatment | weekly for up to 16 weeks
length/height gain during treatment | weekly for up to 16 weeks
changes to phase angle (PhA) as measured by bioelectrical impedance analysis | up to weekly for up to 16 weeks
changes to extracellular water (ECW) as measured by bioelectrical impedance analysis | up to weekly for up to 16 weeks
changes to total body water (TBW) as measured by bioelectrical impedance analysis | up to weekly for up to 16 weeks
changes to fat free mass as measured by bioelectrical impedance analysis | up to weekly for up to 16 weeks
changes in immunological function during treatment as measured by quantification of T-cell recombination excision circles (TRECs) and kappa-deleting recombination excision circles (KRECs) on dried blood spots | up to weekly for up to 16 weeks
rates of acute illness, including diarrhea, vomiting, and fever during treatment | weekly for up to 16 weeks
mortality | up to 16 weeks
hospitalization | up to 16 weeks
duration of treatment required prior to short-term recovery | up to 16 weeks
medium-term vital status | up to 6 months post-recovery
  calculated as number of children who die divided by total number of children initially enrolled
medium-term nutritional status | up to 6 months post-recovery
  calculated as number of children who develop acute malnutrition by the total number of children initially enrolled
medium-term rates of relapse to SAM | up to 6 months post-recovery
medium-term rates of relapse to MAM | up to 6 months post-recovery
medium-term rates of hospitalization | up to 6 months post-recovery
medium-term weight gain | up to 6 months post-recovery
medium-term MUAC gain | up to 6 months post-recovery
medium-term length/height gain | 6 months post-recovery
medium-term phase angle (PhA) as measured by bioelectrical impedance analysis | 6 months post-recovery
medium-term extracellular water (ECW) as measured by bioelectrical impedance analysis | 6 months post-recovery
medium-term total body water (TBW) as measured by bioelectrical impedance analysis | 6 months post-recovery
medium-term fat free mass as measured by bioelectrical impedance analysis | 6 months post-recovery
medium-term immunological function during treatment as measured by quantification of T-cell recombination excision circles (TRECs) and kappa-deleting recombination excision circles (KRECs) on dried blood spots | 6 months post-recovery
short-term cost-efficiency | up to 16 weeks
  calculated as the total costs of the treatment for all children divided by the number of children who achieve nutritional recovery
medium-term cost-efficiency | 6 months post-recovery
  calculated as the total costs of the treatment for all children divided by the number of children who sustain nutritional recovery

CONTACTS AND LOCATIONS:
Overall Officials: Heather C Stobaugh, PhD, Principal Investigator — Action Against Hunger USA; Indi Trehan, MD MPH DTM&H, Principal Investigator — University of Washington; Yosef B Asefaw, MSc, Principal Investigator — Ethiopian Public Health Institute
Locations (3):
- Ethiopia (3):
  - Sekota, Sekota, Amhara
  - Teltele, Teltelē, Oromiya
  - Gode, Gode, Somali

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Trehan I, Beyene Y, Darsene H, Adams BS, Wrabel M, Gizaw G, Legese LA, Cichon B, Chitekwe S, Shellemew MW, Tessema M, Stobaugh HC. The Modified Dosages for Acute Malnutrition (MODAM) study: protocol for three integrated randomized controlled trials of novel approaches for the management of childhood wasting in Ethiopia. BMC Nutr. 2025 Apr 8;11(1):71. doi: 10.1186/s40795-025-01054-w. PMID 40200326